CLINICAL TRIAL: NCT00003620
Title: A PHASE II STUDY OF FLAVOPIRIDOL (NSC # 649890) IN PATIENTS WITH PREVIOUSLY TREATED BCELL CHRONIC LYMPHOCYTIC LEUKEMIA
Brief Title: Flavopiridol in Treating Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02280; CALGB-19805; U10CA031946 (NIH); CDR0000066699 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-09-25 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia; Stage I Chronic Lymphocytic Leukemia; Stage II Chronic Lymphocytic Leukemia; Stage III Chronic Lymphocytic Leukemia; Stage IV Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — alvocidib

ARMS (1):
- Treatment (flavopiridol) (Experimental): Patients registered before 9/15/2000 receive flavopiridol IV continuously on days 1-3. Treatment repeats every 14 days for a total of 12 courses in the absence of disease progression or unacceptable toxicity.
  Patients registered after 9/15/2000 receive flavopiridol IV over 1 hour daily on days 1-3. Treatment repeats every 3 weeks for a total of 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: alvocidib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of flavopiridol in treating patients who have chronic lymphocytic leukemia that has not responded to treatment with fludarabine. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
OBJECTIVES: Determine the complete and partial response rate to flavopiridol in patients with fludarabine-refractory chronic lymphocytic leukemia.

Assess the toxicity profile of this treatment in these patients. Examine progression-free survival and overall survival following this treatment in these patients.

Determine the effects of flavopiridol on normal T-cell subsets and immunoglobulin levels in these patients.

OUTLINE: This is an open label, multicenter study.

Patients registered before 9/15/2000 receive flavopiridol IV continuously on days 1-3. Treatment repeats every 14 days for a total of 12 courses in the absence of disease progression or unacceptable toxicity.

Patients registered after 9/15/2000 receive flavopiridol IV over 1 hour daily on days 1-3. Treatment repeats every 3 weeks for a total of 8 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for the first year and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed intermediate risk (stage I or II) or high risk (stage III or IV) refractory B-cell chronic lymphocytic leukemia
* Intermediate risk group must have evidence of active disease as shown by at least one of the following:

  * Massive or progressive splenomegaly and/or lymphadenopathy
  * Weight loss of greater than 10% in the last 6 months
  * CALGB grade 2-4 fatigue
  * Fevers greater than 100.5 degree Fahrenheit OR night sweats for greater than2 weeks without evidence of infection
  * Progressive lymphocytosis with an increase greater than 50% over a 2 month period or an anticipated doubling time of less than 6 months
* Refractory to fludarabine treatment OR relapsed within 6 months of fludarabine
* Lymphocytosis greater than 5000/mm3 at some time during disease
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Creatinine no greater than 1.5 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No more than 1 prior nonradiolabeled antibody treatment (e.g., Campath-1H or rituximab)
* At least 1, but no more than 3, prior chemotherapy regimens
* At least 1 prior chemotherapy regimen comprising fludarabine
* No other concurrent chemotherapy
* No concurrent chronic use of oral corticosteroids
* No concurrent hormone therapy except for non-disease related conditions
* No concurrent dexamethasone or other corticosteroid-based antiemetics
* No concurrent palliative radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 1999-06; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Complete + partial response rate | Up to 5 years
  The CR + PR rate will be estimated with a 95% confidence interval, and the success of the study will be judged with the two-stage design given above.

SECONDARY OUTCOMES:
Toxicity profile of flavopiridol | Up to 5 years
  Toxicities will be tabulated by type and grade
Progression-free survival | From onstudy date to the date of progression or death, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method.
Overall survival | From onstudy date to the date of death, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: John Byrd, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States